CLINICAL TRIAL: NCT01150604
Title: Depression Management Project (DMP)
Brief Title: Depression Management Project
Acronym: DMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T32MH019391 (NIH)
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Major Depression; Depression
Keywords: Cognitive Behavioral Therapy; Mood Management; Self-help; Internet
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Self-help course (Experimental)
  Interventions: Behavioral: Self-help cognitive-behavioral online course

INTERVENTIONS:
Behavioral: Self-help cognitive-behavioral online course — A self-help online course based on cognitive behavioral therapy for major depression.

SUMMARY:
The purpose of this study is to determine whether an eight-lesson self-help intervention delivered online will result in a reduction of depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 18 years of age or older,
* Participants will have regular (>1 time/week) access to internet and email, with a valid email address,
* Participants will be fluent or almost fluent in English, and
* Participants will be looking for information to help themselves, rather than another person.
* Only those invited to participate will be eligible.

Exclusion Criteria:

* Participants under 18 years of age,
* Participants will with sporadic (< 1 time/week) access to internet and email,
* Participants who fail to provide an email address,
* Participants with English difficulties,
* Participants looking for information to help someone else, and
* Participants not invited will be ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptoms - Self-report | Baseline, 1, 2, and 5 months post consent

CONTACTS AND LOCATIONS:
Overall Officials: Yan Leykin, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States